CLINICAL TRIAL: NCT03282981
Title: Beta Adrenergic Antagonist For The Healing of Chronic Diabetic Foot Ulcers
Brief Title: Beta Adrenergic Antagonist for the Healing of Chronic DFU
Acronym: BAART-DFU
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: VA Northern California Health Care System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SURG-004-16F; 17-08-00792 (Other Grant/Funding Number: VA Northern California Health Care System)
Record Dates: First submitted 2017-09-12; First posted 2017-09-14 (Actual); Results first posted 2025-04-25 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-04

CONDITIONS: Chronic Diabetic Foot Ulcers; Diabetic Neuropathic Ulcers; Non Healing Wound
MeSH Terms: interventions — Timolol; Hydrogels

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Timolol (Experimental): Timoptic-XE plus standard of care (SOC)
  Interventions: Drug: Timolol
- SOC plus non biologically active gel (Placebo Comparator): SOC plus non biologically active gel (hydrogel as placebo medication)
  Interventions: Drug: Non biologically active gel

INTERVENTIONS:
Drug: Timolol — Topical application of Timolol on non-healing diabetic foot ulcers
  Other Names: Timoptic-XE
  Arms: Timolol
Drug: Non biologically active gel — Topical application of non biologically active gel (Hydrogel- standard of care) on non-healing diabetic foot ulcers
  Other Names: Hydrogel
  Arms: SOC plus non biologically active gel

SUMMARY:
One in four Veterans is affected by diabetes and will develop a diabetic foot ulcer. Diabetic ulcers are very challenging to manage and are the most common cause of leg amputation. Many advanced treatments are expensive and difficult to use in the clinic or at home. Those newer therapies have shown little success in healing diabetic foot wounds. The investigators' laboratory and animal work has suggested that a safe medication, currently used as an eye drop for treatment of glaucoma, can heal these ulcers. The investigators are proposing to test this drop (timolol) directly on the surface of the foot ulcer to see if can improve healing faster than the current standard of care. To do this, the investigators propose a "randomized controlled trial" with two groups of patients with diabetic foot ulcers: one will receive standard of care with timolol while the other will receive standard of care with a gel (hydrogel, as placebo medicine).

DETAILED DESCRIPTION:
The trial is designed as a prospective, randomized, double-blinded controlled study of subjects presenting with diabetic foot ulcers. The purpose of this study is to evaluate the superiority of Timoptic-XE therapy in conjunction with standard of care (SOC) treatment (Group A: Timoptic-XE + SOC) versus SOC (Group B: SOC + plus a non-biologically active gel, i.e., hydrogel, as placebo medication) in the clinical effectiveness in promoting wound healing and closure.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject of any race 18 years old or older
* Lower extremity ulcer located anywhere on the foot (as defined as beginning below the malleoli of the ankle):

  * Of more than 30 days duration and less than 2 years duration
  * Surface area between 0.5cm2 and 20cm2 (as measured with the Silhouette imaging system at randomization). The ulcer with largest surface area meeting inclusion criteria will be selected as index ulcer
  * If two ulcers present with the same surface area, the ulcer of the longest duration will be selected as index ulcer
* Documented Ankle Brachial Index (ABI) between 0.8 and 1.2 on the study limb or toe pressure over 65mmHg within 3 months of screening phase
* Documented biopsy report to rule out malignancy of ulcer of > 6 months duration
* Subject or legally authorized representative understands and is willing to give written informed consent
* Subject or legally authorized representative is willing and able to comply with a trial (13 to 17 days) of protocol-specified standard care prior to randomization and to comply with all study requirements

Exclusion Criteria:

* Ulcer of non-diabetic etiology, such as venous, arterial and burn wounds
* Index ulcer is less than 3 cm in distance from any other ulcer on the same extremity
* There are greater than 3 ulcers on the study foot
* Index ulcer presents with any of the following: cellulitis, osteomyelitis, exposed bone, tendon or fascia, capsule , purulent exudate or gangrene
* Index ulcer shows evidence of infection (defined as a moderate or severe rating of all of the following clinical signs/symptoms:

  * increased warmth
  * increased pain
  * erythema
  * malodorous exudate at Screening or at Randomization (Visit 1), OR total organism count > 1 x 105 colony forming units (CFU) from the screening visit study ulcer culture sample)
* Index ulcer surface area has decreased or increased > 40% between Screening and at Randomization (Visit 1) as assessed by the Silhouette imaging system
* Has acquired or is known to be infected with Human Immunodeficiency Virus (HIV)
* Has active malignancy on the study foot
* Has uncontrolled diabetes mellitus as defined by glycosylated hemoglobin A1C > 12%
* Has immunodeficiency as defined by serum IgG, IgA, and IgM less than one-half the lower limit of normal
* Has severe protein malnutrition as defined by serum albumin < 2.5 g/dL
* Has serum aspartate aminotransferase (AST, SGOT, GOT) or serum alanine aminotransferase (ALT, SGPT, GPT) levels greater than twice the upper limit of normal
* Has fatigue, palpitations, dyspnea, and/or angina at rest
* Has a history, within the previous 12 months from date of Screening Visit, of alcohol or drug abuse, particularly methadone or heroin
* Has received previous treatment with the following during the 60 days prior to Screening:

  * Immunosuppressive agents
  * radiation
  * chemotherapy
  * growth factors (epidermal growth factor, tumor necrosis factor, transforming growth factor, platelet derived growth factor, etc.)

    * at the site of the study ulcer, split- or full-thickness skin graft at the site of the study ulcer, biologically-active (or engineered) cellular or acellular product(s) at the site of the study ulcer, investigational drug or device
* Has been hospitalized for treatment of a diabetic foot ulcer within the previous 30 days from Screening
* Has history of heart block 2nd and 3rd degree
* Female who is pregnant or refuses to use adequate contraceptive methods and is of childbearing age during the trial
* Prisoners, institutionalized individuals or vulnerable population

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2018-07-24 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2024-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sara E. Dahle, DPM MPH, Principal Investigator — VA Northern California Health Care System, Mather, CA; Rivkah R. Isseroff, MD, Principal Investigator — VA Northern California Health Care System, Mather, CA
Locations (1):
- VA Northern California Health Care System, Mather, CA, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kaur R, Tchanque-Fossuo C, West K, Hadian Y, Gallegos A, Yoon D, Ismailyan L, Schaefer S, Dahle SE, Isseroff RR. Beta-adrenergic antagonist for the healing of chronic diabetic foot ulcers: study protocol for a prospective, randomized, double-blinded, controlled and parallel-group study. Trials. 2020 Jun 8;21(1):496. doi: 10.1186/s13063-020-04413-z. PMID 32513257

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment started on July 24, 2018 and continued until August 30, 2023 from clinics at the VA Northern California Health Care System.
Period: Overall Study
Arm/Group | Timolol | SOC Plus Non Biologically Active Gel
Started (24 subjected completed study) | 21 | 27
Completed | 21 | 24
Not Completed | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Timolol | SOC Plus Non Biologically Active Gel | Total
Number analyzed (Participants) | 21 | 27 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 68 (8) | 67 (8) | 68 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 20 | 27 | 47
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 5 | 9
  White | 16 | 19 | 35
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 3 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 21 | 27 | 48

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Complete Wound Closure, as Assessed Over a 12 Week Period
Description: Complete wound closure will be assessed by Investigators and is defined as 100% epithelialization of the wound site ("skin re-epithelialization without drainage or dressing requirements by Week 12). The primary outcome was the proportion of patients with complete wound healing by the end of the treatment phase, evaluated using Fisher's exact test.
Time Frame: 12 weeks
Population: chronic, diabetic foot ulcerations
Measure: Count of Participants; unit: Participants
Arm/Group | Timolol | SOC Plus Non Biologically Active Gel
Number analyzed (Participants) | 21 | 27
Participants | 8 | 7

2. Primary Outcome: Safety Outcome Measurement of Timolol Serum
Description: Safety outcome measurement of timolol serum during the treatment phase. Serum Timolol levels were assessed in all participants receiving SOC + Timolol. Most levels were below the detectable limit (<0.22 ng/mL), suggesting minimal systemic absorption. Three participants exhibited detectable levels, with one case of a protocol deviation involving excessive application resulting in a serum level of 1.00 ng/mL. No systemic effects were observed in these cases, supporting the safety profile of topical Timolol.
Time Frame: 12 weeks
Population: safety level measure of serum timolol
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Timolol | SOC Plus Non Biologically Active Gel
Number analyzed (Participants) | 21 | 0
ng/ml | 0.596 (0.315) |

3. Secondary Outcome: The Time to Wound Closure Between the Two Groups
Time Frame: 31 weeks
Population: chronic diabetic foot ulcer
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | Timolol | SOC Plus Non Biologically Active Gel
Number analyzed (Participants) | 21 | 27
weeks | 5.8 (1.0) | 9.2 (1.0)

ADVERSE EVENTS:
Time Frame: 5 years
Arm/Group | Timolol | SOC Plus Non Biologically Active Gel
All-Cause Mortality (participants affected / at risk) | 2/21 | 5/27
Serious Adverse Events (participants affected / at risk) | 0/21 | 2/27
Other Adverse Events (participants affected / at risk) | 0/21 | 0/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Timolol (N=21) | SOC Plus Non Biologically Active Gel (N=27)
Infection (Infections and infestations) | 0 (0) | 1 (1) — Infection
Lightheadedness (Metabolism and nutrition disorders) | 0 (0) | 1 (1) — Lightheadedness

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-07-16): https://cdn.clinicaltrials.gov/large-docs/81/NCT03282981/Prot_SAP_000.pdf